CLINICAL TRIAL: NCT03547219
Title: Biomarkers of Antidepressant Response and Suicidal Events in Depressed Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University (Other)
Collaborators: National Research Foundation of Korea (Other)
Responsible Party: Principal Investigator, Jae-Won Kim, Professor, Seoul National University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2015R1A2A2A01004501
Record Dates: First submitted 2018-05-24; First posted 2018-06-06 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Depression; Adolescent
Keywords: Depression; Adolescent; Biomarker; Inflammation; Brain-derived neurotrophic factor (BDNF); Functional MRI; Antidepressant; Machine learning
MeSH Terms: conditions — Depression; Inflammation | interventions — Escitalopram

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Escitalopram (Experimental): Participants with depression were treated with escitalopram(ranging from 5mg to 30mg) for 8 weeks. Escitalopram was initiated at 5mg for 1 week, followed by an increase to 10mg at week 2. After week 2, doses of escitalopram were titrated according to symptoms and adverse effects. Specific, indicated psychotherapy for depression was not allowed during the study.
  Interventions: Drug: Escitalopram

INTERVENTIONS:
Drug: Escitalopram
  Other Names: Lexapro

SUMMARY:
The aims of this study are to (1) identify inflammatory/neurotrophic and neurodevelopmental markers that predict antidepressant response and suicidal risk in depressed youth and (2) predict their treatment response and the occurrence of suicidal events at the individual level using machine learning approach.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of major depressive disorder(MDD) according to criteria of Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5)
* current episode at least 4 weeks in duration at baseline
* with a score of at least 40 on the Children's Depression Rating Scale-Revised (CDRS-R), and CGI-Severity ≥4 at baseline

Exclusion Criteria:

* intelligence quotient (IQ) lower than 70
* psychotic features or first-degree relatives with a history of bipolar I disorder
* alcohol or substance abuse within the past 6 months
* history of schizophrenia, bipolar disorder, eating disorder, or autism
* history of neurological diseases including convulsive disorders or brain damage
* concurrent medications with psychotropic effects (other than stimulants for ADHD)
* chronic medical conditions (e.g., asthma, inflammatory bowel disease, diabetes) and/or chronic medication with psychotropic effects (e.g., anticonvulsants) or chronic use of NSAIDS or other drugs with known impact on inflammatory pathways.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 152 (Actual)
Dates: Start 2015-08-05 (Actual); Primary Completion 2018-08-02 (Actual); Study Completion 2018-08-02 (Actual)

PRIMARY OUTCOMES:
the change from baseline in CDRS-R at week 8 or upon termination | baseline and 8 weeks or upon termination
  The Children's Depression Rating Scale-Revised (CDRS-R) is a clinician-rated scale to measure the severity of depression of children and adolescents. The CDRS-R consists of 17 items. Depression symptoms are rated on a 5-point scale from 1 to 5 for sleep, appetite, and tempo of speech items and a 7-point scale from 1 to 7 for remaining 14 items. The total score ranges form 17 (normal) to 113 (severe depression).
  Change from baseline CDRS-R at 8 weeks or upon termination was calculated as baseline minus 8 weeks in the adjusted CDRS-R total score (CDRS-R total minus 17, the minimum possible total score).

SECONDARY OUTCOMES:
CGI-I at 8 weeks or upon termination | baseline and 8 weeks or upon termination
  The Clinical Global Impression - Improvement scale (CGI-I) is a 7 point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention. and rated as: 1=very much improved; 2= much improved; 3=minimally improved; 4=no change from baseline; 5=minimally worse; 6=much worse; 7=very much worse since the initiation of treatment.
  CGI-I was measured at 8 weeks or upon termination

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Won Kim, MD, PhD, Principal Investigator — Seoul National University and Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, N/A = Not Applicable, South Korea

REFERENCES:
- [Derived] Choi CH, Lee J, Lee KH, Hong SB, Kim SH, Han JY, Kim JW, Cho SC, Kim JW. Effects of Antidepressant Treatment on Symptom Measures of Attention in Adolescents with Depression: A Preliminary Open-Label Study. J Child Adolesc Psychopharmacol. 2021 May;31(4):288-293. doi: 10.1089/cap.2020.0101. Epub 2021 Jan 8. PMID 33417814